CLINICAL TRIAL: NCT00018447
Title: Combination Osteogenic Therapy in Established Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-022-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Osteoporosis, Post-Menopausal
Keywords: osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Parathyroid Hormone

INTERVENTIONS:
Drug: PTH 1-34
Drug: MFPSR-fluoride

SUMMARY:
This study is designed to determine if combining parathyroid (PTH 1-34) with fluoride (MFPSR) therapy in a cyclic treatment regimen will: (1) produce a greater increase in bone density of the spine than would be produced by either treatment alone; (2) prevent the resistance (i.e., decreased bone formation and no further increase in bone density) that is observed within 18-24 months of PTH therapy; (3) eliminate the calcium deficiency and osteomalacia that can occur with fluoride; (4) prevent excessive bone fluoride content; and (5) result in an increase in bone density which is maintained after treatment is discontinued.

DETAILED DESCRIPTION:
This is a 3-yr, single center, open label, active controlled, randomized study of approximately 99 postmenopausal females with osteoporosis of spine or femoral neck. Patients will be assigned to 1 of 3 groups: 1) PTH 1-34; 2) Fluoride; 3) PTH and fluoride. The treatment period is 3 years with 3-month cycles of therapy. PTH will be administered subcutaneously by injection 600 units daily for 28 days the first month of each 3-month cycle. Fluoride will be administered orally one 76mg tablet twice daily (providing 20 mg fluoride/day), during the last 2 months of each cycle. Calcium will be provided 800mg/day during month 1 and 1500-2000mg for months 2 and 3 of each cycle.

ELIGIBILITY:
* Female, aged 60-80,
* Postmenopausal greater than or equal to 5 years,
* BMD -2.5 to -4.0 at lumbar spine or femoral neck and one standard deviation below young adult mean in the other site, or -2.0 with fracture.
* Vertebral fracture 0-1.

Exclusion Criteria:

* More than 1 vertebral fracture in lumbar spine or more than 4 fracture in the T-L spine.
* Weight less than 45 kg or more than 80 kg, or more than 25% above ideal body weight.
* Present cardiac disease present.
* Diseases or conditions known to affect bone metabolism.
* Therapies with drugs that affect bone metabolism within 6 months.
* Fluoride or Biophosphonates at any time.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Study Completion 2003-10

CONTACTS AND LOCATIONS:
Locations (1):
- Jerry L. Pettis Memorial Veterans Medical Center, Loma Linda, California, United States